CLINICAL TRIAL: NCT04452305
Title: Spermatogonial Stem Cell (SSC) Transplant and Testicular Tissue Grafting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kyle Orwig, Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20030111
Record Dates: First submitted 2020-06-18; First posted 2020-06-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Infertility, Male; Cancer; Autoimmune Disorder
Keywords: spermatogonial stem cells; testis; fertility; oncofertility
MeSH Terms: conditions — Infertility, Male; Neoplasms; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spermatogonial Stem Cell Transplant & Testicular Tissue Graft (Experimental): Stem cell transplantation Testicular tissue grafting
  Interventions: Procedure: Spermatogonial Stem Cell Transplant and Testicular Tissue Grafting

INTERVENTIONS:
Procedure: Spermatogonial Stem Cell Transplant and Testicular Tissue Grafting — Spermatogonial stem cell transplant and testicular tissue grafting is performed to produce sperm.

SUMMARY:
Spermatogonial stem cell transplantation through ultrasound guided rete testis injection and testicular tissue grafting will be performed for participants who have frozen testicular tissue prior to gonadotoxic therapy. The purpose of this study is to test the safety and feasibility of these transplant technologies and restore fertility for these participants.

DETAILED DESCRIPTION:
Azoospermia (no sperm in ejaculated semen) impacts 1% of men in the general population and 15% of infertile men, which translates to 645,000 males between the ages of 20 and 50 (prime reproductive years) in the United States. Spermatogenesis arises from a population of spermatogonial stem cells in the testes that maintain continuous sperm production throughout a man's post-pubertal life. Diseases or medical treatments that compromise the stem cell pool and/or prevent the stem cells from differentiating can cause infertility. Adult men have the option to cryopreserve a semen sample prior to therapy but this is not an option for prepubertal patients who are not yet producing sperm. This study will test the safety and feasibility of two approaches to restore sperm production using previously cryopreserved testicular tissues, which contain spermatogonial stem cells.

The first approach is autologous transplantation of testicular cells, including spermatogonial stem cells, into the testis using ultrasound-guided rete testis injection. The second approach is autologous grafting of intact pieces of testicular tissue under the skin in the scrotum.

ELIGIBILITY:
Inclusion Criteria:

* Male participant at least in Tanner stage 3
* Previously cryopreserved and stored testicular tissue/cells (frozen due to an infertility-risking diagnosis or treatment such as chemotherapy or radiation) available for autologous transplantation and grafting
* Healthy enough to undergo anesthesia
* Written clearance for the procedure from the patient's hematologist or oncologist to confirm the patient has finished treatment for primary condition and are clear to undergo autologous stem cell transplant

Exclusion Criteria:

* Participants considered to be high risk for surgical complications
* Participants with a history of leukemia, lymphoma or testicular cancer or a cancer that likely involved testicles at the time of testicular tissue collection
* Diagnosed with psychological, psychiatric, or other conditions which prevent giving fully informed consent.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with return of spermatogenesis | 3 months-1year
  Rate of participants where sperm was found in semen analysis or testicular tissue analysis

SECONDARY OUTCOMES:
Number of participants with cancer recurrence | 5 years
  Rate of participants diagnosed with cancer recurrence
Number of participants with surgical complications of SSC transplantation and testicular tissue grafting | 3 months
  Rate of infection, hospital readmission, re-operation occurs

CONTACTS AND LOCATIONS:
Overall Officials: Kyle E Orwig, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will publish individual participant data, after deidentification. The investigators will also report each individual participants data back to them. Participants will be identified with unique ID numbers. No identifiable information will be shared.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed at korwig@mwri.magee.edu

REFERENCES:
- [Derived] Zielen AC, Peters KA, Shetty G, Gross DA, Hanna CB, Dovey SL, Wecht A, Cannon GM, Meistrich ML, Hsieh M, Hwang K, Orwig KE. Ultrasound-Guided Rete Testis Approach to Sperm Aspiration and Spermatogonial Stem Cell Transplantation in Patients with Azoospermia. medRxiv [Preprint]. 2025 Mar 26:2025.03.25.25324518. doi: 10.1101/2025.03.25.25324518. PMID 40365444